CLINICAL TRIAL: NCT07195175
Title: First in Human, Randomized, Blinded, Placebo-Controlled Single Ascending Dose and Multiple Dose Study of MAR002 in Healthy Men
Brief Title: Study of MAR002 in Healthy Men
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Marea Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: MAR-201
Record Dates: First submitted 2025-08-27; First posted 2025-09-26 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Acromegaly
MeSH Terms: conditions — Acromegaly

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind (sponsor unblinded), placebo-controlled single ascending dose and multiple dose
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Dose A MAR002 (Experimental): Subcutaneous injection
  Interventions: Drug: MAR002; Drug: Placebo
- Dose B MAR002 (Experimental): Cohort 2 receiving single Dose B
  Interventions: Drug: MAR002; Drug: Placebo
- Dose C MAR002 (Experimental): Cohort 3 receiving single Dose C
  Interventions: Drug: MAR002; Drug: Placebo
- Dose D MAR002 (Experimental): Cohort 4 receiving single Dose D
  Interventions: Drug: MAR002; Drug: Placebo
- Dose E MAR002 (Experimental): Cohort 5 receiving single Dose E
  Interventions: Drug: MAR002; Drug: Placebo
- Dose F MAR002 (Experimental): Cohort 6 receiving multiple Dose F
  Interventions: Drug: MAR002; Drug: Placebo

INTERVENTIONS:
Drug: MAR002 — subcutaneous injection
Drug: Placebo — Subcutaneous injection

SUMMARY:
Evaluate the safety and tolerability of subcutaneous (SC) administration of MAR002 in healthy men

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent
2. Age 18 to 40
3. Weight 55 to 95 kg
4. Body mass index (BMI) 18 to 30 kg/m2
5. Healthy men

Exclusion Criteria:

1. History of hypersensitivity to monoclonal antibodies or study drug
2. Participation in any other investigational drug study
3. History of cancer
4. Recent acute illness
5. Positive test for HIV, hepatitis B/C
6. History of substance abuse or nicotine use
7. Recent blood donation
8. History of pituitary disorder
9. Any condition that prevents the participant from complying with study procedures

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-08-11 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of participants with TEAEs (treatment-emergent adverse events) | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the safety and tolerability of subcutaneous (SC) administration of MAR002 in healthy men

SECONDARY OUTCOMES:
PK Parameters -- Cmax | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (Cmax)
PK Parameters - Tmax | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (Tmax)
PK Parameters - AUC | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (AUC)
PK Parameters - Half Life | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (Half Life)
PK Parameters - Clearance | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (Clearance)
PK Parameters - MRT | From first dose of study drug through final End of Study/Early Termination Visit. End of Study is Day 64 for Cohorts 1 and 2; End of Study is day 169 for Cohorts 3, 4, 5, and 6.
  To evaluate the PK parameters through plasma concentration (MRT)

CONTACTS AND LOCATIONS:
Locations (1):
- Marea Site, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided